CLINICAL TRIAL: NCT03528135
Title: Project PRIDE: Intervention to Reduce HIV Risk in Young Sexual Minority Men
Brief Title: Project PRIDE (Promoting Resilience In Discriminatory Environments)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Houston (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Nathan G. Smith, Associate Professor, University of Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 111889; 1R21DA041250-01A1 (NIH)
Record Dates: First submitted 2018-03-26; First posted 2018-05-17 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Human Immunodeficiency Virus; Sexually Transmitted Infections; Anxiety; Depression; Substance Use Disorders
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Sexually Transmitted Diseases; Anxiety Disorders; Depression; Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: The study includes a randomized controlled trial with one intervention condition and one wait-list control condition. All participants will complete the pre-test and be randomized to receive Project PRIDE immediately or to wait approximately 5 months before receiving it. Randomization will occur as follows: for each recruitment wave (n = 41 per wave), 41 sealed envelopes, each containing a card with the condition (14 cards labeled "wait-list" for the wait-list control group; 27 labeled "group to start shortly" for the intervention group), will be pinned to a foam board. Each participant will choose one card and open it. Those in the intervention group will be assigned to one of two groups of 13-14 participants. After completing the 8 sessions, those in the intervention and those in the matched control will complete the post-test. Approximately 3 months later, these participants will complete the follow-up; those in the control will then receive Project PRIDE.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Project PRIDE (Experimental): Those in the Project PRIDE condition will receive 8 weekly sessions, each lasting 2.5 hours and consisting of approximately 10 men (estimated number given expected attrition). Each session will be co-led by two trained group facilitators. The intervention sessions are described in the "Detailed Description" section. The will complete a pre-test, post-test, and follow-up assessment.
  Interventions: Behavioral: Project PRIDE
- Wait-list (No Intervention): Those in the wait-list arm will wait approximately 5 months before receiving the intervention. They will complete the same pre-test, post-test, and follow-up assessments as those in the PRIDE arm. After they have completed the follow-up assessment, they will be offered the intervention.

INTERVENTIONS:
Behavioral: Project PRIDE — See arms section.
  Arms: Project PRIDE

SUMMARY:
The specific aims are to:

1. Pilot test a randomized controlled trial of Project PRIDE for feasibility for subsequent research projects. A sample of 123 men aged 18-25 who identify as gay, bisexual, queer, or some other non-heterosexual identity, who are HIV negative, who report at least once instance of condomless anal sex in the absence of PrEP in the past 60 days, and who report drug use at least once in the past 60 days will be recruited and randomized to one of two conditions:

   1. Project PRIDE: an eight-session primary HIV-prevention intervention; or
   2. Wait-list control condition: after approximately 5 months, participants will receive Project PRIDE.
2. Test the feasibility of obtaining biological measures of stress, drug use, and HIV/sexually transmitted infection (STI) status. To examine the impact of the intervention on stress physiology, participants will provide saliva samples that will be used to assess diurnal stress (i.e., cortisol) at pre-test, post-test, and 3-month follow-up. To substantiate self-report measures, participants will provide urine samples that will be used to assess drug use. Participants will be tested for gonorrhea, and chlamydia at each time point by providing a separate urine sample, HIV via oral swab and for syphilis by providing a blood sample.
3. It is hypothesized that, compared to the wait-list control group, those in the treatment group will report significant reductions in mental health problems (depression, anxiety. loneliness), minority stressors (internalized homonegativity, sexual orientation concealment), substance use (drug and alcohol), condomless anal sex, number of sex partners, and stress-related biomarkers (salivary cortisol). In addition, compared to the wait-list control group, those in the treatment group will report significant improvements in self-esteem.

DETAILED DESCRIPTION:
Project PRIDE is a manualized group intervention consisting of 8 weekly sessions, each lasting 2.5 hours and consisting of approximately 10 men (estimated number given expected attrition). Each session will be co-led by two trained group facilitators. The intervention sessions will proceed as follows.

Sessions 1 and 2 will consist of introductions, setting of ground rules, exploration of expectations and apprehensions, a broad exploration of participants' different gay/bisexual (GB) identities, and an introduction to the minority stress theory. Special attention will be paid to creating a safe space for all participants and the establishment of a non-judgmental, sex-positive atmosphere.

Sessions 3 and 4 will consist of an introduction to the stress and coping model, application of the model via a group activity to facilitate understanding, and an exploration of GB-associated stressors in different areas of participants' lives (e.g., friendships, romantic and/or sexual relationships, school/work, family). Participants will be asked to set specific mental and behavioral (i.e., sexual and drug use) health goals using the SMART (specific, measurable, attainable, realistic, and time-bound) goal-setting model.

Session 5 will consist of identifying links between sexual behavior, minority stress, and coping, with an emphasis on triggers for sexual risk behavior such as drug use.

In Sessions 6 and 7 safer sexual practices and sexual communication skills will be addressed through group activities and psychoeducation, with an emphasis on harm reduction and normalization. Examples of activities include demonstration of proper condom application using a penis model, demonstration of opening an internal condom, and watching a video regarding the importance of using lubricant during anal sex. An example of sexual communication includes the explanation and demonstration of assertive communication, with an emphasis on assertive communication regarding one's sexual needs and boundaries. Participants will have opportunities for active engagement, such as role-plays to practice assertive communication.

Session 8 will consist of a review of the topics covered in the group and participants' experiences in group, with emphasis on what participants learned and what topics participants thought they still needed to focus on. The group leaders will seek feedback regarding the areas of the intervention that were effective and ineffective. Finally, participants will be given a chance to say goodbye to the leaders and other members.

At pre, post, and follow-up, participants will complete self-report questionnaires, containing a demographic questionnaire and the measures listed in section 9. Participants will complete all measures on a password-protected laptop computer. In addition, participants will complete urine drug tests and tests for HIV, chlamydia, gonorrhea, and syphilis. Finally, participants will collect their saliva at four time points at each assessment to assess for cortisol awakening response.

ELIGIBILITY:
Inclusion Criteria:

* Self-identification as male
* Self-identification as gay, bisexual, queer, or some other non-heterosexual identity
* Aged 18-25
* HIV-negative as assessed via OraQuick
* Self-report of at least one instance of condomless anal or vaginal sex (insertive or receptive) while not taking Truvada for pre-exposure prophylaxis (PrEP) in the past 60 days
* Self-report of drug use in the past 60 days
* Willingness to complete HIV/STI test, drug test, questionnaires, and randomization
* Willingness to collect and return saliva
* Ability and willingness to stop prescription medication on the day of saliva collection
* Proficient in English

Exclusion Criteria:

* Failure to meet any inclusion criterion will result in exclusion from the study

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Participants who self-identify as male (regardless of sex assigned at birth) are eligible.
Enrollment: 17 (Actual)
Dates: Start 2018-11-09 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Change in 60-Day Condomless Anal Sex in the Absence of PrEP from pre-test to 5 months | Pre-test, approximately 2 months after pre-test, approximately 5 months after pre-test
  Frequency of condomless anal sex in the absence of pre-exposure prophylaxis (i.e., use of Truvada to prevent HIV) will be assessed using the Timeline Followback method (Robinson, Sobell, Sobell, & Leo, 2014), a calendar-based method for assessing the type and frequency of sexual contact and is sensitive to changes over time. This measure will be administered separately from the other measures, using an Excel document. Each participant will complete a 60-day Timeline Followback for sexual behaviors.

SECONDARY OUTCOMES:
Salivary cortisol | Pre-test, approximately 2 months after pre-test, approximately 5 months after pre-test
  Salivary cortisol will be completed by all participants who will be provided with kits and detailed oral and written instructions for proper saliva collection to measure diurnal cortisol. Participants will collect their saliva at pre, post, and follow-up. Participants will collect saliva (1) upon awakening, (2) 30 minutes after awakening and prior to brushing teeth, (3) 90 minutes after awakening, and (4) before going to bed and note collection times in writing. Samples 1-3 are required as an assessment of the cortisol awaking response (CAR). Sample 4 represents a potential lower-limit because hormone levels are typically down-regulated to a low-point prior to going to sleep. Participants will be instructed to avoid eating, drinking beverages other than water, smoking, or chewing gum 30 minutes before saliva collection.
60-Day Drug Use | Pre-test, approximately 2 months after pre-test, approximately 5 months after pre-test
  All HIV-negative participants will provide a urine sample for toxicology, using the RapidCheck 9 Multi-Drug Test Panel to validate self-reports and assess drugs used. The RapidCheck 9 Multi-Drug Test Panel is a rapid, one-step diagnostic test that screens for nine targeted illicit and prescription drugs and their metabolites at the minimum cutoff sensitivity levels established by the National Institute on Drug Abuse. The nine targeted drugs are tetrahydrocannabinol (THC), Cocaine, phencyclidine (PCP), Opiates, Methamphetamine including Ecstasy, Methadone, Amphetamines, Barbiturates, and Benzodiazepines. Urine samples will be collected at Avenue 360. Study personnel will complete the testing of urine using the RapidCheck 9 Multi-Drug Test Panel at Avenue 360. The results of the RapidCheck 9 will be entered into an online survey hosted by Qualtrics with the participant's study identification (ID) number. Urine will be discarded after testing and will not leave Avenue 360.
60-Day Self-Reported Drug/Alcohol Use | Pre-test, approximately 2 months after pre-test, approximately 5 months after pre-test
  Self-reported drug/alcohol use will be assessed using the Timeline Followback method (Robinson, Sobell, Sobell, & Leo, 2014), a calendar-based method for assessing drug and alcohol use frequency and amount that is sensitive to changes in use. This measure will be administered separately from the other measures, using an Excel document. Each participant will complete a 60-day Timeline Followback for alcohol use, cocaine/crack, and methamphetamines. Each Excel document will be saved on the password-protected University of Houston laptop and identified by the participant study ID.
Loneliness | Pre-test, approximately 2 months after pre-test, approximately 5 months after pre-test
  Loneliness will be measured using the UCLA Loneliness Scale (Russell, 1996), a 20-item scale that measures experiences of loneliness. Cronbach alphas ranged from .89 to .94.
Self Esteem | Pre-test, approximately 2 months after pre-test, approximately 5 months after pre-test
  Self esteem will be measured by the Rosenberg Self-esteem Scale (Rosenberg, 1965), a 10-item scale that measures feelings of self worth. Cronbach alpha was .87.
Coping | Pre-test, approximately 2 months after pre-test, approximately 5 months after pre-test
  Coping will be measured using the Ways of Coping Questionnaire (WOC) (S. Folkman & Lazarus, 1988), a 66-item measure that assesses the degree to which participants use certain coping strategies to deal with a stressor. Cronbach alphas ranged from .61 to .79.
Racist Discrimination | Pre-test, approximately 2 months after pre-test, approximately 5 months after pre-test
  Racist discrimination will be measured among ethnic/racial minority participants only using the Racial Microaggressions Scale (Torres-Harding, Andrade Jr, & Romero Diaz, 2012), a 32-item measure of racist invalidations. Cronbach alpha ranged from .78 to .89.
Anti-Gay/Bisexual Discrimination | Pre-test, approximately 2 months after pre-test, approximately 5 months after pre-test
  Anti-GB discrimination will be measured by the Heterosexist Harassment, Rejection, and Discrimination Scale (Szymanski, 2006), a 14-item scale that measures experiences of sexual orientation-based discrimination. Cronbach alphas ranged from .74 to .89.
Gay/Bisexual Identity | Pre-test, approximately 2 months after pre-test, approximately 5 months after pre-test
  Gay/bisexual identity will be measured by the Lesbian, Gay, and Bisexual Identity Scale (Mohr & Kendra, 2011), a 27-item scale that measures facets of gay and bisexual identity. Cronbach's alpha ranged from .76 to .89
Internalized Homonegativity | Pre-test, approximately 2 months after pre-test, approximately 5 months after pre-test
  Internalized homonegativity will be measured by the Nungesser Homosexuality Attitudes Inventory-Revised (Nungesser, 1983), a 36-item scale measuring negative attitudes towards one's own homosexuality. Cronbach alpha was .94.
Anxiety | Pre-test, approximately 2 months after pre-test, approximately 5 months after pre-test
  Anxiety will be measured using the state version of the State-Trait Inventory for Cognitive and Somatic Anxiety (Grös, Antony, Simms, & McCabe, 2007), a 21-item scale measuring cognitive and somatic symptoms of anxiety. Cronbach alpha was .92.
Depression | Pre-test, approximately 2 months after pre-test, approximately 5 months after pre-test
  Depression will be measured using the Center for Epidemiologic Studies Depression Scale (Radloff, 1977), a 20-item scale measuring depressive symptoms. Cronbach alphas ranged from .84 to .90.
HIV | Pre-test, approximately 5 months after pre-test
  All participants will be screened for HIV (rapid OraQuick test) with pre- and post-test counseling. Pre-test counseling will include a description of the test and meaning of test results, discussion of possible responses to positive results, the possible consequences of disclosing HIV information, and legal protections against unauthorized disclosure. Post-test counseling will include the results and discussion of their meaning, referrals for treatment if indicated, and a review of risk-reduction strategies. The pre- and post-test counseling protocol will follow the State of Texas Health Department protocols and will be in adherence with Texas laws governing HIV testing and confidentiality. HIV/STI testing and pre- and post-test counseling will be administered by trained staff at Avenue 360. In addition to referral to treatment, those testing positive for HIV will be excluded from the study.
Gonorrhea | Pre-test, approximately 2 months after pre-test, approximately 5 months after pre-test
  All participants will be tested for gonorrhea (via urine test) with pre- and post-test counseling. Pre-test counseling will include a description of the tests and meaning of test results, discussion of possible responses to positive results, the possible consequences of disclosing STI information, and legal protections against unauthorized disclosure. Post-test counseling will include the results and discussion of their meaning, referrals for treatment if indicated, and a review of risk-reduction strategies. The pre- and post-test counseling protocol will follow the State of Texas Health Department protocols and will be in adherence with Texas laws governing STI testing and confidentiality. STI testing and pre- and post-test counseling will be administered by trained staff at Avenue 360.
Chlamydia | Pre-test, approximately 2 months after pre-test, approximately 5 months after pre-test
  All participants will be tested for chlamydia (via urine test) with pre- and post-test counseling. Pre-test counseling will include a description of the tests and meaning of test results, discussion of possible responses to positive results, the possible consequences of disclosing STI information, and legal protections against unauthorized disclosure. Post-test counseling will include the results and discussion of their meaning, referrals for treatment if indicated, and a review of risk-reduction strategies. The pre- and post-test counseling protocol will follow the State of Texas Health Department protocols and will be in adherence with Texas laws governing STI testing and confidentiality. STI testing and pre- and post-test counseling will be administered by trained staff at Avenue 360.
Syphilis | Pre-test, approximately 2 months after pre-test, approximately 5 months after pre-test
  All participants will be tested for syphilis (via blood test) with pre- and post-test counseling. Pre-test counseling will include a description of the tests and meaning of test results, discussion of possible responses to positive results, the possible consequences of disclosing STI information, and legal protections against unauthorized disclosure. Post-test counseling will include the results and discussion of their meaning, referrals for treatment if indicated, and a review of risk-reduction strategies. The pre- and post-test counseling protocol will follow the State of Texas Health Department protocols and will be in adherence with Texas laws governing STI testing and confidentiality. STI testing and pre- and post-test counseling will be administered by trained staff at Avenue 360.
60-Day Vaginal Sex | Pre-test, approximately 2 months after pre-test, approximately 5 months after pre-test
  Vaginal sex frequency will be assessed using the Timeline Followback method (Robinson, Sobell, Sobell, & Leo, 2014), a calendar-based method for assessing the type and frequency of sexual contact and is sensitive to changes over time. This measure will be administered separately from the other measures, using an Excel document. Each participant will complete a 60-day Timeline Followback for sexual behaviors.
60-Day Oral Sex | Pre-test, approximately 2 months after pre-test, approximately 5 months after pre-test
  Oral sex frequency will be assessed using the Timeline Followback method (Robinson, Sobell, Sobell, & Leo, 2014), a calendar-based method for assessing the type and frequency of sexual contact and is sensitive to changes over time. This measure will be administered separately from the other measures, using an Excel document. Each participant will complete a 60-day Timeline Followback for sexual behaviors.

CONTACTS AND LOCATIONS:
Overall Officials: Nathan G Smith, PhD, Principal Investigator — University of Houston
Locations (1):
- Avenue 360, University of Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Smith NG, Hart TA, Kidwai A, Vernon JRG, Blais M, Adam B. Results of a Pilot Study to Ameliorate Psychological and Behavioral Outcomes of Minority Stress Among Young Gay and Bisexual Men. Behav Ther. 2017 Sep;48(5):664-677. doi: 10.1016/j.beth.2017.03.005. Epub 2017 Apr 4. PMID 28711116
- [Background] Smith NG, Hart TA, Moody C, Willis AC, Andersen MA, Blais M, Adam B. Project PRIDE: A cognitive-behavioral group intervention to reduce HIV risk behaviors among HIV-negative young gay and bisexual men. Cognitive and Behavioral Practice 23:398-411, 2016.